CLINICAL TRIAL: NCT05966285
Title: Suture Repair vs Mesh Repair in the Treatment of Incarcerated Groin Hernia in Elderly Populations: a Retrospective, Single-center Study
Brief Title: Suture Repair vs Mesh Repair in the Treatment of Incarcerated Groin Hernia in Elderly Populations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: Huadong Hospital to FDU
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Incarcerated Groin Hernia
Keywords: Incarcerated groin hernia; Emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- suture group: Patients ≥65 years who underwent urgent surgical groin hernia repair from January 2015 to June 2022 were included.
  Interventions: Other: suture repair
- mesh repair: Patients ≥65 years who underwent urgent surgical groin hernia repair from January 2015 to June 2022 were included.
  Interventions: Other: mesh repair

INTERVENTIONS:
Other: suture repair — Suture repair was used to reinforce the abdominal wall, including Bassini, Ferguson, McVay, or Halsted technique.
  Groups: suture group
Other: mesh repair — Mesh repair was conducted using a synthetic and biological mesh in the Lichtenstein or open preperitoneal techniques.
  Groups: mesh repair

SUMMARY:
Purpose:

Tension-free hernia repair is the gold standard for groin hernia repair. However, there is no consensus on the optimal surgical treatment for incarcerated groin hernia in elderly populations, The aim of this study was to compare the clinical efficacy of mesh repair and suture repair in the treatment of incarcerated groin hernia in elderly patients.

Methods:

Patients ≥65 years who underwent urgent surgical groin hernia repair from January 2015 to June 2022 will be included. Patient demographic data and short-term and long-term postoperative outcomes will be retrospectively analyzed.

DETAILED DESCRIPTION:
This study includes consecutive patients ≥65 years diagnosed with IGH who underwent emergency surgical repair at our center between January 2015 and June 2022. The study is conducted in compliance with the ethical standards laid down in the 1964 Declaration of Helsinki and its subsequent amendments.

Only true emergencies were included in the study, involving IGH patients who underwent urgent surgical repair within six hours of an emergency admission or patients who underwent emergency surgery due to sudden exacerbation while awaiting elective repair surgery during hospitalization. Various techniques were performed to repair IGH during the surgical procedure. In cases where there was no ischemic necrosis of the hernia contents, the hernia content was simply reduced, followed by high ligation of the hernia sac at the inner ring of the groin. Subsequently, mesh repair was conducted using a synthetic and biological mesh in the Lichtenstein or open preperitoneal techniques, while suture repair was utilized in the Bassini, Ferguson, or Halsted operation. For femoral hernias, McVay repair was used in suture repair while open preperitoneal techniques was used for mesh repair. In cases of IGH accompanied by intestinal necrosis, the initial procedure involved resection of the necrotic bowel followed by in vitro anastomosis through a groin incision. Subsequently, high ligation of the hernia sac was carried out, and the choice between mesh or tissue repair was left to the discretion of the surgeon. The choice of surgical techniques was based on the surgeons' experience and the overall condition of the patient. Based on the surgical method used, the researchers were categorized into two groups: suture repair and mesh repair groups.

After hospital discharge, the patient was scheduled for regular outpatient visits for at least 1 year of follow-up, physical Examination and patient's subjective perceptions were used to determine the presence of recurrence or other long-term complications. The end of the follow-up was June 2023. Recorded death, recurrence, or loss to follow-up were considered to be the endpoint.

Investigators collected data on the following three aspects: (1) patients' demographic information, including age, sex, American Society of Anesthesiologists (ASA) grade, previous abdominal operation, previous surgical repair of groin hernia, history of acute incarceration, comorbidities, and time from incarceration to surgery; (2) surgical details, such as the type of groin hernia, preoperative antibiotic use, nighttime surgery (the start time of surgery was from 5 p.m. to before 8 a.m. the next day), hernia contents, bowel resection, hernia sac size, area of the hernia ring, prosthetic material used, open or laparoscopic surgery, type of anesthesia (general anesthesia or spinal anesthesia), placement of the drainage; and (3) clinical outcomes, which included postoperative recurrence as a long-term outcome, and the surgery related death, surgical site infection (SSI) within 30 days, length of hospital stay, ICU admission, and overall wound complications as short-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with incarcerated groin hernia (IGH).
2. Aged ≥65 years
3. Received emergency surgical repair (mesh or suture repair) at our center between January 2015 and June 2022.

Exclusion Criteria:

* IGH patients did not undergo either mesh repair or suture repair.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥65 years diagnosed with incarcerated groin hernia (IGH) who underwent emergency surgical repair.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Recurrence | at least one year
  Recurrence is determined by physical examination or the patient's subjective perceptions

SECONDARY OUTCOMES:
length of hospital stay | up to 3 months
  The number of days from hospitalization to discharge
length of ICU stay | up to 3 months
  The number of days in ICU
surgery-related death | within 30 days after surgery
  Deaths occurring during the first hospital stay
surgical site infection | within 30 days after surgery
  would infection
overall complications | at least 1 months
  combination of Outcome 1 to 6

IPD SHARING:
Plan to Share IPD: No